CLINICAL TRIAL: NCT04325139
Title: External Validation of a Predictive Model for Bowel Preparation in Patients Undergoing Colonoscopy
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: KT20200324-3
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Bowel Preparation; Colonoscopy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Before colonoscopy, the following information was obtained by the colonoscopists through asking patients: the characteristics of last stool, the time of drinking first dose of laxative, the time of first defecation, the time of drinking last dose of laxative. The beginning time of colonoscopy was also recorded. During withdrawal phase, the quality of bowel preparation was evaluated based on BBPS scale.

SUMMARY:
Bowel preparation is closely lined to the quality of colonoscopy, inadequate bowel preparation (IBP) could lead to higher miss rate of adenomas, patients' discomfort and higher health expense. For the patients with possible IBP before the examination, it may be better to cancel the colonoscopy and repeat bowel preparation through modified or enhanced strategies. This study aimed to externally validate the efficiency of a procedure-based model in predicting inadequate bowel preparation

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Patient undergoing colonoscopy

Exclusion Criteria:

* Patients with prior colectomy
* Unable to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study involving eleven tertiary-centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation | 1 hour
  Defined by each segmental BBPS≥2

SECONDARY OUTCOMES:
The rate of yellow, clear stool in the last defecation | 1 hour
  The characteristics of the last stool was self-evaluated by patients based on a picture containing different kind of stool examples.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Department of Gastroenterology, Hongai Hospital, Xiamen, Fujian
  - Xiang'an hospital of Xiamen University, Xiamen, Fujian
  - Department of Gastroenterology, Qionghai people's hospital, Qionghai, Hainan
  - Department of Gastroenterology, Bethune international peace hospital, Shijiazhuang, Hebei
  - Department of Gastroenterology，Zhengzhou Central Hospital, Zhengzhou, Henan
  - Department of Gastroenterology, Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shannxi
  - Department of Gastroenterology，Shanxi Bethune hospital, Taiyuan, Shanxi
  - Department of Gastroenterology，Chengdu third people's hospital, Chengdu, Sichuang
  - Department of Gastroenterology, The First Affiliated Hospital of the Medical College, Shihezi University, Shihezi, Xinjiang